CLINICAL TRIAL: NCT02968303
Title: Phase 2 Study With COmbination of Vemurafenib With Cobimetinib in B-RAF V600E/K Mutated Melanoma Patients to Normalize LDH and Optimize Nivolumab and Ipilimumab therapY
Brief Title: Induction Therapy With Vemurafenib and Cobimetinib to Optimize Nivolumab and Ipilimumab Therapy
Acronym: COWBOY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Isala (Other)
Responsible Party: Principal Investigator, Rutger Koornstra, Medical Oncologist, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOMEL27 - COWBOY
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Melanoma, Malignant, of Soft Parts
MeSH Terms: conditions — Sarcoma, Clear Cell | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction treatment (Experimental): Induction vemurafenib and cobimetinib (6 weeks) directly followed by ipilimumab and nivolumab
  Interventions: Drug: Vemurafenib and Cobimetinib
- No induction treatment (No Intervention): Upfront ipilimumab and nivolumab without induction by vemurafenib and cobimetinib

INTERVENTIONS:
Drug: Vemurafenib and Cobimetinib — Combination of Vemurafenib with Cobimetinib in BRAF V600E/K mutated melanoma patients to normalize LDH and optimize immunotherapy with Nivolumab and Ipilimumab
  Arms: Induction treatment

SUMMARY:
Rationale:

The combination of ipilimumab and nivolumab induces relatively high response rates and promising response depth in late stage melanoma. Nevertheless, it takes time till responses occur and still a significant number of patients do not benefit from treatment, due to rapid progressive disease or resistance to therapy.

In contrast to immunotherapies targeted therapies (BRAF or MEK inhibitors), can induce faster and higher response rates, but often of shorter duration, even when combined.

Initial attempts of combining vemurafenib or dabrafenib + trametinib with ipilimumab failed due to toxicity.

Patients with elevated levels of serum LDH are less likely to respond to immunotherapy compared to patients with normal LDH levels. This does not mean that such patients do not benefit at all from immunotherapy.

This raises the question, whether response rates upon immunotherapy can be improved by upfront reduction of tumor burden and normalization of LDH.

The investigators postulate that induction therapy with combined BRAF+MEK inhibition, and subsequent LDH normalization, can improve response rates to the rates seen in LDH normal patients.

To address this question the investigators have setup a randomized phase 2 trial in metastatic melanoma patients with elevated serum LDH comparing the response rates upon ipilimumab + nivolumab versus ipilimumab + nivolumab preceded by 6 weeks of vemurafenib + cobimetinib induction.

Furthermore, less than half of the patients treated with the combination of ipilimumab and nivolumab received maintenance nivolumab, and approximately 40% of all patients discontinued treatment for toxicity. In 70% of patients responses were ongoing despite discontinuation of treatment due to toxicity. This raises the question, to what extent does maintenance therapy add clinical benefit to an ongoing immune response. Preclinical data indicate even that continuous restimulation of T cells can result in activation induced non-responsiveness (anergy).

Therefore, a secondary objective of this trial will be, to test a response-driven nivolumab scheme

Objectives:

Primary Objective • To compare efficacy of induction vemurafenib + cobimetinib followed by ipilimumab + nivolumab (Arm A) versus upfront ipilimumab + nivolumab treatment (Arm B).

Secondary Objectives

* To describe duration of response and overall survival induced by vemurafenib + cobimetinib followed by the combination of ipilimumab + nivolumab (Arm A) as compared to ipilimumab + nivolumab (Arm B)
* To describe the rate and quality of toxicity observed in the two study arms
* To describe the rate of ongoing responses upon response-driven flat dose (240mg q2w or 480mg q4w) nivolumab maintenance
* To determine the immune-activating capacity of induction therapy with vemurafenib + cobimetinib followed by the combination of ipilimumab + nivolumab.
* To evaluate the changes in systemic immune competence

Study design:

This is a two-arm phase 2 study consisting of 200 BRAFV600E/K mutation-positive late-stage melanoma patients with an elevated baseline LDH level (> ULN, < 3xULN) randomized 1:1 (stratified according to LDH) to receive either vemurafenib + cobimetinib directly followed by ipilimumab + nivolumab (Arm A) or standard first line ipilimumab + nivolumab (Arm B). Subsequently, patients in both arms will receive flat dose (240mg q2w or 480mg q4w) nivolumab maintenance in a response-driven manner.

Study population:

Stage IV, or unresectable stage III, BRAFV600E/K mutation positive melanoma patients, naïve for BRAF/MEK, PD-1/PD-L1 or CTLA-4 targeting therapy, 18 years and older.

Intervention:

Patients will be randomized 1:1 to receive either 6 weeks vemurafenib 960 mg bid + cobimetinib 60 mg QD 21-day on, 7-day off (21/7) schedule, directly followed by 4 courses of ipilimumab 3mg/kg q3wk + nivolumab 1mg/kg q3wk (Arm A) or first line standard 4 courses of ipilimumab 3mg/kg q3wk + nivolumab 1mg/kg q3wk (Arm B).

Subsequently, patients in both arms will receive nivolumab maintenance flat dose (240mg q2w or 480mg q4w) in a response-driven manner according to their response at week 18.

Main study parameters/endpoints:

Primary Endpoints

• Compare the best overall response rate (BORR) according to RECIST 1.1 of both arms at week 18 from start of treatment.

Secondary Endpoints

* Progression-free survival (PFS) according to RECIST 1.1
* Overall survival (OS)
* Percentage of grade 3/4 toxicities according to CTCv4.03
* Percentage of ongoing response, percentage of patients requiring re-induction, response percentage upon re-induction
* Changes in tumor-specific T cell responses

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* World Health Organization (WHO) Performance Status 0-2
* Histologically or cytologically confirmed Stage IV, or unresectable stage III, BRAF V600E/K mutated melanoma
* Measurable disease according to RECIST 1.1
* Signed and dated informed consent form
* No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1
* No prior BRAFi and/ or MEKi therapy
* No immunosuppressive medications
* Screening laboratory values must meet the following criteria and should be obtained within 10 days prior to randomization:

  * WBC ≥ 2.0x109/L, Neutrophils ≥ 1.0x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 5.0 mmol/L
  * Creatinine ≤ 2x ULN or creatinine clearance (CrCl) ≥ 40 ml/min
  * AST, ALT ≤ 3.0 x ULN (≤5 x ULN for patients with liver metastases)
  * Bilirubin ≤ 2.0 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL )
  * LDH > ULN, < 5.0 x ULN
* No symptomatic brain metastases (asysmptomatic brain metastases, accidentally found during screening can be included)
* No leptomeningeal metastases
* No active autoimmune disease requiring systemic treatment in the past 3 months or a documented history of autoimmune disease, or history of syndrome that required systemic steroids, at daily dose of ≥10mg prednisone or equivalent, or immunosuppressive medications. (Subjects with vitiligo or resolved childhood asthma/atopy are excluded from this rule (and will not be excluded from this study). Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.)
* No evidence of interstitial lung disease or active, non-infectious pneumonitis
* No active infection requiring therapy
* No known additional malignancy that is progressing or requires active treatment
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days + the time required for nivolumab to undergo five half-lives) after the last dose of study medication
* WOBCP must have a negative serum or urine pregnancy test within 96 hours prior to the start of study treatment and must not be breast feeding
* Men must agree to the use of male contraception during the study treatment period and for at least 31 weeks after the last dose of study drug.
* Currently not participating in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* No underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Best overall response rate (BORR) according to RECIST 1.1 | Week 18 from start of treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) according to RECIST 1.1 | 1 and 2 years from start of treatment
Overall survival (OS) | 1 and 2 years from start of treatment
Grade 3/4 toxicities according to CTCv4.03 | Week 18 from start of treatment
Percentage of ongoing response | 1 and 2 years from start of treatment
Response percentage upon re-induction | Week 18 from start of treatment
Changes in tumor-specific T cell responses | Week 18 from start of treatment

CONTACTS AND LOCATIONS:
Locations (13):
- Netherlands (13):
  - The Netherlands Cancer Institute, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis Breda, Breda
  - Maxima MC, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum Heerlen, Heerlen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht UMC+, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided